CLINICAL TRIAL: NCT03862326
Title: The Effect of Group-, Individual-, and Ultrasound Guided Pelvic Floor Training on Incontinence
Brief Title: Pilot Study - Patient Education and Pelvic Strength Exercises in Elderly Women With Incontinence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg Municipality (Other)
Responsible Party: Principal Investigator, Signe Refsgaard Bech, Pricipal Investigator, University College of Northern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-20160049
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 3 arms, one with group exercises, one with individual exercises and one with ), Individual exercises guided by ultrasonography imaging
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and outcome assessor did not know what treatment the indivdual women got.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Training (Other): Group Training of the women with incontinence - with 5-8 women in each group. This is also Usual Care
  Interventions: Behavioral: Exercise
- Individual training (Experimental): Individual pelvic floor exercises one-to-one with the physiotherapist
  Interventions: Behavioral: Exercise
- Individual training with biofeedback (Experimental): Individual pelvic floor exercises one-to-one with the physiotherapist but with ultrasound used as biofeedback, and to check if the women are contracting the right muscles.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — From lying to sitting to active exercises with focus on the pelvic floor
  Other Names: Behaviour

SUMMARY:
It will be investigate if women with a diaper grant in Aalborg Municipality can reduce diaper size and thus costs for diapers in the municipality through meetings with a incontinence nurse and pelvic floor exercises.

DETAILED DESCRIPTION:
Incontinence is a world wide challenge especially in elderly women. The participation in pelvic floor exercises can to some extent help women with urinary incontinency. In the Municipality of Aalborg in Denmark, the citizens can get a diaper grant, if they are incontinence. The project will be recruiting women with diaper grants and randomly allocate the women to 3 different groups 1) Group training (usual care), 2) Individual training and 3) Individual training with biofeedback in the form of ultrasound. All groups will receive the same incontinence education from the incontinence nurses and physiotherapists. The Women will be offered 6 individual or 10 group base trainings, with increased time between trainings, to increase the participants independency and rely more on home based exercises.

ELIGIBILITY:
Inclusion Criteria:

Diaper grant

* Urinary incontinency Living in own home in Aalborg Municipality

Exclusion Criteria:

* Dementia Inability to transport herself to the training facility neurological diseases inability to understand Danish or bring a translator

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Pelvic floor strength | Change compared to baseline after 12 week intervention
  Change in pelvic floor strength measured through internal palpation with the use of oxford Scale (0-5, where 5 is the highest strength) but transferred to percentage and normalized to baseline values.
Pelvic floor strength | Change compared to baseline 3 months after end of intervention.
  Change in pelvic floor strength measured through internal palpation with the use of oxford Scale (0-5, where 5 is the highest strength) but transferred to percentage and normalized to baseline values.

SECONDARY OUTCOMES:
Change in life quality - UDI-6 | after 12 weeks of exercise and 3 months follow-up
  Urinary Distress Inventory (UDI-6) questionnaire with a total score, in each of the 6 questions the subjects scores between 0 to 3, 0 being Not at all, 1 being A little bit, 2 being Moderately and 3 being Greatly
Change in life quality IIQ-7 | after 12 weeks of exercise and 3 months follow-up
  Incontinence Impact Questionnaire (IIQ-7) questionnaire with a total score, in each of the 7 questions the subjects can score between 0 to 3, 0 being Not at all, 1 being A little bit, 2 being Moderately and 3 being Greatly

CONTACTS AND LOCATIONS:
Overall Officials: Signe R Bech, Phd, Principal Investigator — University College of Northern Denmark
Locations (1):
- Signe Refsgaard Bech, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322